CLINICAL TRIAL: NCT02367612
Title: Fermented Milk on the Appearance of Common Winter Infectious Diseases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 210/12ES1
Record Dates: First submitted 2015-02-12; First posted 2015-02-20 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Acute Gastroenteritis; Upper Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Cultured Milk Products

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fermented milk (Experimental): Fermented milk with Lactobacillus paracasei CBA L74
  Interventions: Dietary Supplement: Fermented milk
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Fermented milk — Fermented milk with Lactobacillus paracasei CBA L74
  Arms: Fermented milk
Dietary Supplement: Placebo — Maltodextrin
  Arms: Placebo

SUMMARY:
Respiratory and gastrointestinal infections are common in children under the age of 4 years, especially after the start of schooling. These conditions are facilitated by a still incomplete functional maturation of the immune system and the anatomical structure and function of the respiratory and gastrointestinal tract still developing. The frequency and duration of these conditions involves a high discomfort and significant costs, in relation to medical appointments, taking medication, the need for hospitalization, days of absence from school and work days lost by parents. Functional foods derived from the fermentation of cow's milk with probiotic strains have been proposed for the prevention of infectious diseases in children. Several products have been investigated, with sometimes conflicting results. Diversity in experimental designs, populations evaluated, and bacterial strains used in the preparation of fermented products are probably responsible for these discrepancies. Recently we started a study approved by the Ethics Committee for Biomedical Activities "Carlo Romano" of the University of Naples "Federico II" (protocol number 210/12) to evaluate the effectiveness of foods fermented with Lactobacillus paracasei CBA-L74 in the prevention of common winter infections in school children aged between 12 and 48 months. Studies of pre-clinical phase showed anti-inflammatory activity of milk fermented with the strain Lactobacillus paracasei L74-CBA in terms of stimulation of the production of the cytokine IL-10 and decreased synthesis of IL-12, also in response to stimulation with Salmonella typhimurium. The data were obtained in in vitro studies on dendritic cells and ex vivo intestinal biopsies as well as in tests on healthy mice and on a mouse model of experimental colitis. A preliminary analysis of the data was found that subjects treated with fermented milk showed fewer infectious episodes, as well as a lower incidence of respiratory tract infections or gastrointestinal, with a statistically significant difference between the study groups. It was also observed a significant increase in the levels of α- and β- defensins, LL-37 and secretory IgA in the group of subjects treated with fermented milk compared to subjects treated with fermented rice or placebo.

Therefore, we decided to extend the period of study of five additional months, in order to perform an evaluation of the effectiveness of fermented milk (which was more effective)vs placebo.

ELIGIBILITY:
Inclusion Criteria:

* children aged 12-48 months attending educational program (either at nursery or primary school)

Exclusion Criteria:

* concomitant chronic/congenital diseases and disabilities
* active tubercolosis
* congenital cardiac defects
* autoimmune diseases
* immunodeficiency
* cystic fibrosis
* metabolic diseases
* malignancy

  .chronic pulmonary diseases
* malformation of he GI tract
* food allergy
* antibiotic use
* pre/pro/symbiotic use
* severe wasting (less than 3 standard deviations of weight-for-height z score)

Ages: 12 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2014-12; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The occurrence of common winter infectious diseases involving respiratory and/or gastrointestinal tract | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Berni Canani, MD, PhD, Study Director — Federico II University
Locations (3):
- Italy (3):
  - university of naples federico II, Naples, Naples
  - Fabio Mosca, Milan
  - Giovanni Corsello, Palermo